CLINICAL TRIAL: NCT02112864
Title: Impact of Dexamethasone on the Post Operative Inflammatory Response and on the Occurrence of Post Thoracotomy Pain Syndrome
Brief Title: Dexamethasone for Reduction of Post Thoracotomy Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, M.D., M.Sc., Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: dexaPTPS
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain; Dexamethasone; Thoracic Surgery; Cytokines
MeSH Terms: conditions — Chronic Pain | interventions — Dexamethasone; Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone 10 mg (Experimental): Dexamethasone 10 mg will be given as a single-dose, pre incision, intravenously
  Interventions: Drug: Dexamethasone
- normal saline (Placebo Comparator): Patients in this group will receive 2.5 mL of normal saline intravenously, pre-incision
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexamethasone — 10 mg (2.5 ml)
  Other Names: decadron
  Arms: dexamethasone 10 mg
Drug: Normal Saline — 2.5 mL normal saline
  Other Names: Placebo
  Arms: normal saline

SUMMARY:
Post thoracotomy pain syndrome still affects 50% of patients after a thoracic surgery. Pathogenesis is unclear but there is growing evidence that neuro inflammation may play a significant role. Dexamethasone is a very potent anti-inflammatory drug. The hypothesis of this study is that dexamethasone, given pre operatively, would help reduce the incidence of post thoracotomy pain syndrome 3 months after surgery, by reducing the inflammatory response, in patients undergoing elective thoracic surgery that includes thoracic epidural analgesia.

ELIGIBILITY:
Inclusion Criteria:

* elective thoracic surgery using a thoracotomy incision and thoracic epidural analgesia
* ASA I-III
* age 18-75 yo

Exclusion Criteria:

* contra-indication to thoracic epidural analgesia
* patient refusal
* patients already taking cortisone or dexamethasone
* patients on chronic opioid medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-05; Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
cytokine elevation | 24 h after surgery

SECONDARY OUTCOMES:
incidence of post thoracotomy pain syndrome | 3 months after surgery
incidence of post thoracotomy pain syndrome | 6 months after surgery
incisional and shoulder pain | acute post operative period
Brief pain inventory questionnaire | three months after surgery
Brief pain inventory questionnaire | 6 months after surgery
Leeds Assessment of Neuropathic Signs and Symptoms questionnaire | three and six months after surgery
cytokine elevation | 1h after surgery
cytokine elevation | 48 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Brulotte, MD, Msc, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes